CLINICAL TRIAL: NCT05552326
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study of Olezarsen (ISIS 678354) Administered Subcutaneously to Patients With Severe Hypertriglyceridemia
Brief Title: A Study of Olezarsen Administered Subcutaneously to Participants With Severe Hypertriglyceridemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISIS 678354-CS6; 2022-501420-20 (EudraCT Number)
Expanded Access: NCT06360237 (Approved for marketing)
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Severe Hypertriglyceridemia
Keywords: Hypertriglyceridemia; Hyperlipidemias; Metabolic Diseases
MeSH Terms: conditions — Hypertriglyceridemia; Hyperlipidemias; Metabolic Diseases | interventions — olezarsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olezarsen (Experimental): Olezarsen will be administered once every 4 weeks by subcutaneous (SC) injection from Week 1 through Week 49.
  Interventions: Drug: Olezarsen
- Placebo (Placebo Comparator): Olezarsen-matching placebo will be administered once every 4 weeks by subcutaneous (SC) injection from Week 1 through Week 49.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olezarsen — Olezarsen will be administered by SC injection.
  Other Names: ISIS 678354; AKCEA-APOCIII-LRx
  Arms: Olezarsen
Drug: Placebo — Olezarsen-matching placebo will be administered by SC injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of olezarsen as compared to placebo on the percent change in fasting triglycerides (TG) from baseline.

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, randomized, double-blind, placebo-controlled study in 446 participants. Participants will be randomized to receive olezarsen or placebo in a 53-week treatment period. The length of participation in the study will be approximately 78 weeks, which includes an up to 12-week screening period, a 53-week treatment period, and a 13-week post-treatment evaluation period or transition to open-label extension (OLE) study with up to 1-year treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Fasting TG ≥ 500 mg/dL (5.65 mmol/L) at Screening and Qualification
2. Participants must be on lipid-lowering therapy that should adhere to standard of care (SOC) per local guidelines. Lipid-lowering medications should be optimized and stabilized for at least 4 weeks prior to screening to minimize changes in these medications during the study.
3. Participants must be willing to comply with diet and lifestyle recommendations as able.

Exclusion Criteria:

1. Hemoglobin A1c (HbA1c) ≥ 9.5% at Screening
2. Alanine aminotransferase or aspartate aminotransferase > 3.0 × upper limit of normal
3. Total bilirubin > 1.5 ULN unless due to Gilbert's syndrome
4. Estimated GFR < 30 mL/min/1.73 m^2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Fasting TG Compared to Placebo | Baseline and Month 6

SECONDARY OUTCOMES:
Percent Change from Baseline in Fasting TG Compared to Placebo | Baseline and Month 12
Percent Change from Baseline in Fasting Apolipoprotein C-III (ApoC-III), Remnant Cholesterol and Fasting Non-High-Density Lipoprotein-Cholesterol (Non-HDL-C) Compared to Placebo | Baseline, Month 6 and 12
Proportion of Patients Who Achieve Fasting TG <500 mg/dL (5.65 mmol/L) Compared to Placebo | Month 12
Proportion of Participants Who Achieve Fasting TG < 880 mg/dL (10 mmol/L) Compared to Placebo in the Subgroup of Participants with Baseline TG ≥ 880 mg/dL | Month 12
Adjudicated Acute Pancreatitis Event Rate During the Treatment Period Compared to Placebo | Week 1 through Week 53
Absolute Change in Hepatic Fat Fraction (HFF) Between Olezarsen Treatment Group and Pooled Placebo | Baseline through Month 12

CONTACTS AND LOCATIONS:
Locations (204):
- United States (62):
  - Central Research Associates, Inc., Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC Alabaster, Birmingham, Alabama
  - Onyx Clinical Research, Peoria, Arizona
  - NRC Research Institute, Los Angeles, California
  - Accel Research Sites, DeLand, Florida
  - Finlay Medical Research, Greenacres City, Florida
  - University of Florida Jacksonville, Jacksonville, Florida
  - Meridien Research, Maitland, Florida
  - Columbus Clinical Services, Miami, Florida
  - Harmony Clinical Research, Inc, North Miami Beach, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - 3Sync Research, Sunrise, Florida
  - R & B Medical Center LLC, Tampa, Florida
  - JSV Clinical Research Study, Inc., Tampa, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Accel Clinical Research, Eatonton, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Randomize Now, Newnan, Georgia
  - St. Vincent Medical Group, Carmel, Indiana
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Louisville Metabolic and Atherosclerosis Research Center (L-MARC), Louisville, Kentucky
  - Grace Research, LLC, Bossier City, Louisiana
  - Clinical Trials of America LA, LLC, Monroe, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Onyx Clinical Research, Flint, Michigan
  - Onyx Clinical Research, Rochester Hills, Michigan
  - Stern Cardiovascular, Southaven, Mississippi
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Orchard Park Family Practice, Orchard Park, New York
  - Clinical Trials of America, LLC, Lenoir, North Carolina
  - Diabetes and Endocrinology Consultants, P.C., Morehead City, North Carolina
  - OnSite Clinical Solutions, LLC, Salisbury, North Carolina
  - The Ohio State University (OSU), Columbus, Ohio
  - SV Research LLC, Marion, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Main Street Physicians Care Waterway, Little River, South Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - The Jackson Clinic, Jackson, Tennessee
  - Texas Health Family Care, Fort Worth, Texas
  - Vilo Research Group, Houston, Texas
  - Juno Research, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Pioneer Research Solutions, Inc, Houston, Texas
  - Sante Clinical Research, LLC, Kerrville, Texas
  - FMC Science, Lampasas, Texas
  - DCT - McAllen Primary Care, LLC, McAllen, Texas
  - Texas Institute of Cardiology, McKinney, Texas
  - SMS Clinical Research, LLC, Mesquite, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Permian Research Foundation, Odessa, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - Tranquil Research, Webster, Texas
  - Aspen Clinical Research, Orem, Utah
  - Ogden Clinic Grandview, Roy, Utah
  - Clinical Investigation Specialists Inc., Kenosha, Wisconsin
- Argentina (8):
  - CIPREC - Centro de Investigación y Prevención Cardiovascular, Buenos Aires
  - Fundacion Favaloro, Buenos Aires
  - Centro Médico Dra. Laura Maffei, Buenos Aires
  - Glenny Corp SA, Buenos Aires
  - Instituto de Cardiología Corrientes, Corrientes
  - Instituto Médico DAMIC, Córdoba
  - Centro Medico San Luis, San Luis
  - Clínica FUSAVIM Privada, Villa María
- Belgium (4):
  - AZ Sint-Jan Brugge, Bruges
  - Hôpital Erasme, Brussels
  - Virga Jessa Hospital, Hasselt
  - UZ Leuven, Leuven
- Brazil (9):
  - NUPEC - Nucleo de Pesquisa Clinica, Belo Horizonte
  - Núcleo de Pesquisa Clínica, Curitiba
  - Hospital Universitario Walter Cantidio - UFC, Fortaleza
  - Nucleo de Pesquisa em Cirurgia Vascular, Porto Alegre
  - IBPClin Pesquisa Clinica, Rio de Janeiro
  - CPQuali Pesquisa Clinica, São Paulo
  - Instituto do Coração - HCFMUSP, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo - FMUSP, São Paulo
  - i9 Pesquisas Clínicas/Loema - Instituto de Pesquisas Clínica & Consultores, São Paulo
- Bulgaria (16):
  - Medical Center Diamedical EOOD, Dimitrovgrad
  - MHAT Haskovo AD, Haskovo
  - MHAT Pazardzhik AD, Pazardzhik
  - UMHAT - Kaspela EOOD, Plovdiv
  - University Multiprofile Hospital for Active Treatment Pulmed OOD, Plovdiv
  - UMHAT Kanev AD, Rousse
  - MHAT Sliven to MMA Sofia, Sliven
  - Medical Center Smolyan Clinical Research OOD, Smolyan
  - Medical Center for Specialized Medical Help in Cardiovascular Diseases OOD, Sofia
  - Acibadem City Clinic Tokuda University Hospital, Sofia
  - Medico Dental Center ISUL Tsaritsa Yoanna EOOD, Sofia
  - Medical Centre Synexus Sofia EOOD, Sofia
  - Medical Center Zara - Med, Stara Zagora
  - DCC Equita, Varna
  - Specialized Hospital for Active Treatment of Cardiology, Varna
  - Medical Centre "Nevromedics" EOOD, Veliko Tarnovo
- Canada (6):
  - NL Health Services, St. John's, Newfoundland and Labrador
  - Aggarwal and Associates Ltd., Brampton, Ontario
  - Joanne F. Liutkus Medicine Professional Corporation, Cambridge, Ontario
  - Bluewater Clinical Research Group, Sarnia, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Unite de Recherche Clinique, Saint-Jérôme, Quebec
- Czechia (6):
  - CTC Hodonin s.r.o., Hodonín
  - KardioBusak s.r.o., Louny
  - Fakultni nemocnice v Motole, Prague
  - Endokrinologie Cerny Most s.r.o., Prague
  - Diabetologická a endokrinologická ambulance Milan Kvapil, Příbram
  - AeskuLab k.s, Teplice
- France (3):
  - Hopital de Hautepierre, Strasbourg
  - ELSAN - Polyclinique Vauban, Valenciennes
  - GHM les Portes du Sud, Vénissieux
- Greece (5):
  - University General Hospital of Alexandroupoli, Alexandroupoli
  - AHEPA Building of Evaggelismos, Athens
  - University General Hospital ATTIKON, Athens
  - Hygeia Hospital, Athens
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
- Hungary (6):
  - Lausmed Kft., Baja
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - Obudai Egeszsegugyi Centrum, Budapest
  - Clinexpert Kft., Budapest
  - Pharma4 Trial Kft., Gyöngyös
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz Diabetologiai szakrendeles, Kaposvár
- India (10):
  - Max Super Specialty Hospital, New Delhi, National Capital Territory of Delhi
  - B. M. Birla Heart Research Centre A Unit of the Calcutta Medical Research Institute, Kolkata, West Bengal
  - Sri Jayadeva Institute of Cardiovascular Sciences and Research, Bengaluru
  - Sir Ganga Ram Hospital, Delhi
  - Eternal Hospital, Jaipur
  - IPGMER, Kolkata
  - Vinaya Hospital and Research Centre (A Unit of Karnataka Institute of Medical Sciences), Mangaluru
  - KEM Hospital, Mumbai
  - Bhatia Hospital, Mumbai
  - Manipal Hospital Mysore, Mysore
- Italy (4):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - AORN S. Anna e S. Sebastiano UOC FARMACIA, Caserta
  - Azienda Ospedaliero-Universitaria di Ferrara-Arcispedale Sant'Anna, Cona
  - Fondazione I.R.C.C.S. Policlinico "San Matteo" c/o C.U.R.M., Pavia
- Lithuania (5):
  - Saules seimons medicinos centras, Kaunas
  - Klinikiniai sprendimai, Kaunas
  - Clinic of Cardiology and Rehabilitation, Klaipėda
  - Republican Panevezys Hospital, Panevezys
  - Pirmoji viltis, Šiauliai
- Malaysia (4):
  - Sultanah Bahiyah Hospital, Alor Star, Kedah
  - Hospital Taiping, Taiping, Perak
  - Pulau Pinang Hospital, George Town, Pulau Pinang
  - University Malaya Medical Centre (UMMC), Kuala Lumpur
- Mexico (5):
  - Medical Care and Research S.A de C.V., Mérida, Yucatán
  - Centro de Investigación Cardiométabolica de Aguascalientes S.A. de C.V., Aguascalientes
  - Cientia Investigacion Clinica Sc, Chihuahua City
  - Clinstile, S.A. de C.V., Mexico City
  - Clinical Research Institute S.C., Tlanepantla
- Netherlands (7):
  - Vumc Amsterdam Medical Center, Amsterdam
  - Gelre Ziekenhuizen Apeldoorn, Apeldoorn
  - Reinier de Graaf Ziekenhuis, Delft
  - Het Van Weel Bethesda ziekenhuis, Dirksland
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Bethesda Diabetes Research Center, Hoogeveen
  - Canisius-Wilhelmina Ziekenhuis (CWZ), Nijmegen
- Poland (11):
  - UCK, I Klinika Kardiologii, Gdansk
  - Biokinetica, Józefów
  - Centrum Medyczne Pratia, Katowice
  - Centra Medyczne Medyceusz, Lodz
  - Clinical Best Solutions, Lublin
  - Etg Lublin, Lublin
  - Centrum Zdrowia Metabolicznego, Poznan
  - Clinical Best Solutions Sp. Z.o.o Spolka Komandytowa, Warsaw
  - Centrum Medycnze AMED, Warsaw
  - Narodowy Instytut Kardiologii im. S. Wyszyńskiego - PIB, Warsaw
  - ETG Zamosc / Pro Life Medica Sp. z o.o., Zamość
- Portugal (2):
  - Hospital CUF Tejo, Lisbon
  - Centro Hospitalar de Entre Douro e Vouga, Santa Maria da Feira
- Romania (7):
  - Cabinet Medical Individual SC DIANA BARBONTA SRL, Alba
  - Cardioplus Center SRL, Baia Mare
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed S.R.L, Brasov
  - Centrul Medical Medicover Victoria, Bucharest
  - S.C. SAL MED S.R.L., Cardiologie, Piteşti
  - Cardio Med SRL, Târgu Mureş
  - S.C. Mediab Srl, Târgu Mureş
- Slovakia (6):
  - Alian s.r.o., Bardejov
  - Ambulancia diabetologicka a poruch latkovej premeny a vyzivy, Bratislava
  - Interna a diabetologicka ambulancia - IN-DIA s.r.o., Lučenec
  - Diab sro, Rožňava
  - Interna SK, s.r.o., Svidník
  - Areteus s.r.o, Trebišov
- Spain (11):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Comarcal Infanta Elena, Huelva
  - Hospital Universitario de Jaen, Jaén
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional de Malaga, Málaga
  - Unidad de Ensayos Clinicos, Málaga
  - Hospital Provincial de Conxo, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Acardo MedSite, Solna, Sweden
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH), Kaohsiung City
  - Mackay Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/

REFERENCES:
- [Derived] Marston NA, Bergmark BA, Alexander VJ, Prohaska TA, Kang YM, Moura FA, Zimerman A, Waldman E, Weinland J, Murphy SA, Goodrich EL, Zhang S, Xia S, Li D, Goldberg AC, Goudev A, Badimon L, Kiss RG, Vrablik M, Gaudet D, Moulin P, Stroes ESG, Banach M, Cohen H, Blom D, Charng MJ, Nordestgaard BG, Nicholls SJ, Tsimikas S, Giugliano RP, Sabatine MS; CORE-TIMI 72a and CORE2-TIMI 72b Investigators. Olezarsen for Managing Severe Hypertriglyceridemia and Pancreatitis Risk. N Engl J Med. 2026 Jan 29;394(5):429-441. doi: 10.1056/NEJMoa2512761. Epub 2025 Nov 8. PMID 41211918
- [Derived] Marston NA, Bergmark BA, Alexander VJ, Karwatowska-Prokopczuk E, Kang YM, Moura FA, Prohaska TA, Zimerman A, Zhang S, Murphy SA, Tsimikas S, Giugliano RP, Sabatine MS. Design and rationale of the CORE-TIMI 72a and CORE2-TIMI 72b trials of olezarsen in patients with severe hypertriglyceridemia. Am Heart J. 2025 Aug;286:125-135. doi: 10.1016/j.ahj.2025.03.003. Epub 2025 Mar 9. PMID 40064331